CLINICAL TRIAL: NCT05400577
Title: Neoadjuvant Sotorasib in KRAS G12C Mutated, Resectable, Stage Ib-IIIA Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Sotorasib in KRAS G12C Mutated, Resectable, Stage Ib-IIIA NSCLC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Grantor withdrew support due to slow accrual
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-180
Record Dates: First submitted 2022-04-29; First posted 2022-06-01 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sotorasib, 960 mg, oral daily dose for 4 weeks (28 days) (Experimental)
  Interventions: Drug: Sotorasib, 960 mg, oral daily dose for 4 weeks (28 days)

INTERVENTIONS:
Drug: Sotorasib, 960 mg, oral daily dose for 4 weeks (28 days) — Sotorasib, 960 mg, oral daily dose for 4 weeks (28 days)

SUMMARY:
This is a single arm study, conducted at two centers, of neoadjuvant sotorasib in treatment naïve patients with stage Ib-IIIa NSCLC. The study will accrue 25 patients in all. Patients must have been deemed surgically resectable and physiologically fit for surgery by a thoracic surgeon prior to enrollment.

DETAILED DESCRIPTION:
There will be a two-part consent, including consent for KRAS testing and consent for treatment on trial. Testing for a KRAS G12C mutation in patients with resectable, stage Ib-IIIa NSCLC is currently not standard of care. Patients who are otherwise felt to be good candidates for this study, after review in multidisciplinary thoracic tumor board, will be screened for KRAS G12C after signing informed consent for screening. Next generation sequencing will be performed on standard of care diagnostic biopsy tissue for EGFR (standard of care) as well as KRAS mutations. Patients who are found to have a KRAS G12C mutation, will be eligible for the study intervention.

This is a single arm study, conducted at two centers, of neoadjuvant sotorasib in treatment naïve patients with stage Ib-IIIa NSCLC. The study will accrue 25 patients in all. Patients must have been deemed surgically resectable and physiologically fit for surgery by a thoracic surgeon prior to enrollment. In addition, every patient will be discussed in multidisciplinary thoracic tumor board prior to enrollment, with medical oncology, radiation oncology and surgical oncology physicians present, to determine the optimal treatment approach. All patients must undergo baseline tumor staging, including pretreatment biopsy, pathological evaluation of mediastinal lymph nodes (if indicated) by means of bronchoscopy or mediastinoscopy, chest and brain imaging (CT chest with contrast and CT head with contrast or MRI brain); PET and diagnostic CT chest will be repeated within 7 days before surgery. Subjects will take sotorasib dosed at 960 mg daily by mouth with or without food for 4 weeks (28 days) prior to surgery. Changes in tumor size will be evaluated by Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. The primary objective of this study is to determine the rate of MPR. Primary tumors will be assessed, using the recently published International Association for the Study of Lung Cancer guidelines, for percentage of residual viable tumor identified on routine hematoxylin and eosin (H&E) staining, and tumor with no more than 10% viable tumor cells will be considered to have a MPR.

Once patients have completed neoadjuvant therapy, they will undergo surgery, followed by standard of care adjuvant therapy as deemed fit by their treating physician. Data on disease assessment during patients' standard of care visits post-surgery will be collected to evaluate their DFS. All patients will be accrued in 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have non-squamous NSCLC with KRAS G12C mutation identified through molecular testing (local assessment), AJCC 8 stages Ib, IIa, IIb, IIIa (single nodal station) and assessment by a thoracic surgeon that the patient is potentially resectable and physiologically operable. Lymph nodes should be pathologically staged, if feasible, prior to enrollment.
2. No prior NSCLC anticancer therapy
3. Must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v. 1.1 as described in detail in section 11.0.
4. Age > 18 years.
5. ECOG performance status 0 or 1
6. Must have the ability to take oral medications and willing to record daily adherence to investigational product utilizing a sponsor-provided dosing diary
7. Subjects must have normal organ and marrow function as defined below

   * Absolute neutrophil count > 1,000/mcL
   * Platelets > 75,000/mcL
   * Total bilirubin < 1.5 x ULN (< 2.0 x ULN for subjects with documented Gilbert's syndrome or < 3.0 x ULN for whom the indirect bilirubin level suggests an extrahepatic source of elevation)
   * AST/ALT (SGOT/SGPT) < 2.5 times institutional normal limits
   * Creatinine clearance Estimated glomerular filtration rate based on MDRD (Modification of Diet in Renal Disease) calculation >=30 ml/min/1.73 m2
   * Prothrombin time (PT) or partial thromboplastin time (PTT) < 1.5 x ULN, OR International normalized ratio (INR) <1.5 or within target range if on anticoagulation therapy
8. Ability to understand and willingness to sign a written informed consent and HIPAA consent document

Exclusion Criteria:

1. Any prior therapy directed at NSCLC and Previous treatment with a direct KRAS G12C inhibitor.
2. Patients receiving any other investigational agents.
3. Patients with uncontrolled intercurrent illness, that would in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, informed consent, procedures, primary endpoint or study completion. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Patients with non-invasive malignancies (e.g. in situ cervical cancer) ARE eligible.
4. History of allergic reactions attributed to compound of similar chemical or biologic composition to the agent used in this study.
5. Patients receiving any medications or substances that are strong inhibitors or inducers of sotorasib ineligible. Please refer to section 5.2 for details about excluded therapies and restrictions.
6. Major surgery (as assessed by treating clinician) within 28 days of study registration.
7. Pregnant or breast feeding. Refer to section 4.4 for further detail.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response | 2 months
  Major pathologic response is defined as a resection specimen with < or = to 10% viable tumor cells in patients treated with neoadjuvant sotorasib for KRAS G12C mutated, stage Ib-IIIa NSCLC

SECONDARY OUTCOMES:
Determine the safety, feasibility and tolerability of neoadjuvant sotorasib therapy in patients with surgically resectable KRAS G12C mutant NSCLC | 1 months
  Safety is assessed by all treatment-emergent adverse events and treatment-related adverse events. All adverse events will be assessed by the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Borghaei, DO, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No